CLINICAL TRIAL: NCT04537247
Title: A Comparative Study Between Open and Robotic Partial Nephrectomy in Treatment of High Complex Renal Tumors.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Alaa, Assistant lecturer of Urology surgery., Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: open versus robotic PN
Record Dates: First submitted 2020-08-29; First posted 2020-09-03 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-01

CONDITIONS: Renal Tumor
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Open partial nephrectomy (Group A) (Experimental): patients in this group will have open partial nephrectomy for their renal tumors.
  Interventions: Procedure: partial nephrectomy for complex renal tumor
- Robotic partial nephrectomy (group B) (Experimental): patients in this group will have robotic partial nephrectomy for their renal tumors.
  Interventions: Procedure: partial nephrectomy for complex renal tumor

INTERVENTIONS:
Procedure: partial nephrectomy for complex renal tumor — removal of tumor with sufficient safety margin with preservation of functioning renal unit (renal tissue with its collecting system, arterial supply and venous as well as lymphatic drainage).

SUMMARY:
To compare safety and efficacy between open and robotic partial nephrectomy in treatment of organ confined complex renal tumors (R.E.N.A.L score more than 7) as regarding surgical results, morbidity, clinical as well as oncological and functional outcomes.

DETAILED DESCRIPTION:
Although radical nephrectomy was considered as the only effective treatment for malignant kidney tumors and maintained the prime solution for such tumors throughout the nineteenth century, partial nephrectomy became the preferred method in managing tumors of solitary kidneys, bilateral or hereditary renal tumors and in renal tumors of renal insufficiency patients. The shift to preserve sufficient as well as functioning renal volume, the improving experience with renal vasculature, proliferation of energy sources that achieved sufficient tissue cleavage and haemostatic power and refinements in hypothermia techniques helped the shift towards nephron sparing surgeries. Partial nephrectomy aimed at achieving complete removal of renal tumor with preservation of renal function, minimizing ischemia time as well as operative complications.

Open partial nephrectomy was the standard management strategy for organ-confined renal tumors in many centers worldwide. It is still the preferred method in most situations of complex tumors. Yet, open surgery has the inherent problem of poorly cosmetic scar, the need for analgesics, long hospital stay and wound related complications.

Laparoscopic partial nephrectomy (LPN) has largely replaced open partial nephrectomy worldwide as it combines the benefits of nephron sparing surgery (preserving the renal function) and laparoscopy (decreasing morbidity). The increasing experience of LPN enabled surgeons to operate not only small, peripheral, exophytic renal tumors, but also larger infiltrating tumors have been managed similarly. On the other hand, LPN still has technical difficulties that need steep learning curve to be mastered.

Robotic partial nephrectomy has become the surgery of choice not only for most renal tumors but also for benign kidney lesions. The minimally invasive nature of robotic surgery offers numerous advantages to the patient over open surgery including minimal tissue trauma, smaller scars, and faster recovery. Unlike laparoscopy, robotic surgeries grantee a three-dimensional view. The complex operative steps can be easily done due to the wider range of motion of the surgical instruments that the robot provides. Moreover, recent studies showed that robotic partial nephrectomy has shorter ischemia time, less blood loss and faster recovery than laparoscopy.

Despite the multiplicity of studies done for comparing between open and robotic partial nephrectomy in cases of small renal tumors, there are fewer studies comparing between open and robotic partial nephrectomy in management of complex renal tumors, which are not based on randomized bases.

Assiut University Hospitals are intending to be in a leading position in the field of minimal invasive surgery by constructing the first robotic surgery center in Upper Egypt. So, in our study, although robotic surgery seems to be more expensive, investigators suppose that robotic partial nephrectomy will yield better surgical and functional results than open partial nephrectomy in managing complex renal tumors. The promising technology will lead to decrease the robotic industry cost which, till now, remains the major drawback of robotic surgery worldwide spread. Another priority of our intended study is that it will alleviate any selection bias between the two techniques by being a prospective randomized one.

ELIGIBILITY:
Inclusion Criteria:

* Any patient aged more than 18 years old with high complex renal tumor according to R.E.N.A.L scoring system (R.E.N.A.L score more than 7).

Exclusion Criteria:

* 1- Renal tumors with R.E.N.A.L score less than 7, based on radio-logical findings.

  2- Renal tumors in congenitally anomalous kidney (horseshoe kidney, ectopic or malformed) or metastatic kidney disease.

  3- Gross lymphadenopathy (N1 According to TNM classification system of renal tumors) or suspicious vascular invasion (T3a, T3b or T3c according to TNM classification of renal tumors) (18).

  4- Renal pelvic tumor of upper urinary tract. 5- Patient refused to be enrolled in the study. 6- Defaulters of follow up. 7- Bleeding tendency. 8- Active peritoneal or bowel inflammatory process. 9- Clinically unfit patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Successful excision of the tumor. | two years
  Achieving successful excision of the tumor in both open and robotic partial nephrectomy without any operative or immediate post-operative complications.

SECONDARY OUTCOMES:
Status of recurrence free. | two years follow up.
  Patient is free from recurrent tumor in both study groups.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Kamel, M.A urology, Principal Investigator — Faculty of Medicine, Assiut University, Egypt
Locations (1):
- Assiut Urology Hospital, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pavan N, Derweesh IH, Mir CM, Novara G, Hampton LJ, Ferro M, Perdona S, Parekh DJ, Porpiglia F, Autorino R. Outcomes of Laparoscopic and Robotic Partial Nephrectomy for Large (>4 Cm) Kidney Tumors: Systematic Review and Meta-Analysis. Ann Surg Oncol. 2017 Aug;24(8):2420-2428. doi: 10.1245/s10434-017-5831-5. Epub 2017 Mar 16. PMID 28303428
- [Background] Alemozaffar M, Chang SL, Kacker R, Sun M, DeWolf WC, Wagner AA. Comparing costs of robotic, laparoscopic, and open partial nephrectomy. J Endourol. 2013 May;27(5):560-5. doi: 10.1089/end.2012.0462. Epub 2013 Jan 30. PMID 23130756
- [Background] Boylu U, Basatac C, Yildirim U, Onol FF, Gumus E. Comparison of surgical, functional, and oncological outcomes of open and robot-assisted partial nephrectomy. J Minim Access Surg. 2015 Jan-Mar;11(1):72-7. doi: 10.4103/0972-9941.147699. PMID 25598603
- [Background] Wu Z, Li M, Qu L, Ye H, Liu B, Yang Q, Sheng J, Xiao L, Lv C, Yang B, Gao X, Gao X, Xu C, Hou J, Sun Y, Wang L. A propensity-score matched comparison of perioperative and early renal functional outcomes of robotic versus open partial nephrectomy. PLoS One. 2014 Apr 7;9(4):e94195. doi: 10.1371/journal.pone.0094195. eCollection 2014. PMID 24710511
- [Background] Minervini A, Vittori G, Antonelli A, Celia A, Crivellaro S, Dente D, Di Santo V, Frea B, Gacci M, Gritti A, Masieri L, Morlacco A, Porreca A, Rocco B, Parma P, Simeone C, Zaramella S, Carini M, Serni S. Open versus robotic-assisted partial nephrectomy: a multicenter comparison study of perioperative results and complications. World J Urol. 2014 Feb;32(1):287-93. doi: 10.1007/s00345-013-1136-x. Epub 2013 Aug 4. PMID 23913095
- [Background] Wang Y, Shao J, Ma X, Du Q, Gong H, Zhang X. Robotic and open partial nephrectomy for complex renal tumors: a matched-pair comparison with a long-term follow-up. World J Urol. 2017 Jan;35(1):73-80. doi: 10.1007/s00345-016-1849-8. Epub 2016 May 19. PMID 27194142
- [Background] Kim JK, Lee H, Oh JJ, Lee S, Hong SK, Lee SE, Byun SS. Comparison of robotic and open partial nephrectomy for highly complex renal tumors (RENAL nephrometry score >/=10). PLoS One. 2019 Jan 10;14(1):e0210413. doi: 10.1371/journal.pone.0210413. eCollection 2019. PMID 30629644